CLINICAL TRIAL: NCT05276622
Title: Patient and Care Partner Experiences Living With Multiple Myeloma (PaCE-MM)
Acronym: PaCE-MM
Status: Terminated | Type: Observational
Why Stopped: Investigator left the institution.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC2121; 1R03AG074030-01 (NIH)
Record Dates: First submitted 2022-01-26; First posted 2022-03-11 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma
Keywords: Newly diagnosed multiple myeloma; Physical Function; Cognitive Function; Quality of Life; Geriatric Assessments; Care partners
MeSH Terms: conditions — Multiple Myeloma | interventions — Geriatric Assessment; Functional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with newly diagnosed multiple myeloma: Forty subjects with newly diagnosed multiple myeloma.
  Interventions: Other: Comprehensive Geriatric Assessment
- Care partners of the subjects with newly diagnosed multiple myeloma: Thirty care partners of the subjects with newly diagnosed multiple myeloma.
  Interventions: Other: Qualitative patient-care partner interviews; Other: Surveys on well-being and function

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment — A modified Cancer and Aging Research Group (CARG) Geriatric Assessment that includes validated measures of 7 geriatric domains: functional status, comorbidity, cognition, psychological state, social activity, and support, nutritional status, and medications will be performed at baseline (pre-treatment), every 3 months for a total of 3 assessments. The modified comprehensive Geriatric Assessment includes patient-reported surveys and research staff assessments.
  Cognitive Testing: The National Institutes of Health Toolbox Cognition Battery (objective) and PROMIS Short Form v2.0 - Cognitive function 8a (subjective)
  Groups: Subjects with newly diagnosed multiple myeloma
Other: Qualitative patient-care partner interviews — Semi-structured Interviews: Baseline and again at 3 months.
  Groups: Care partners of the subjects with newly diagnosed multiple myeloma
Other: Surveys on well-being and function — Care partner's Surveys on well-being and function: Baseline and again at 3 months
  Groups: Care partners of the subjects with newly diagnosed multiple myeloma

SUMMARY:
This research study is explore the impact over time of multiple myeloma and its associated treatments on the physical and cognitive function and quality of life of patients and their care partners and how these impacts affect the overall illness experience.

DETAILED DESCRIPTION:
This study aims to identify the factors, for example, age, race, sex, education, household income, clinical or other geriatric conditions such as depression, anxiety, or lack of social support that can predict those most likely to experience changes in physical and cognitive function and quality of life. Furthermore, patients and care partners experienced challenges, because of multiple myeloma and its associated treatments, will be studied using semi-structured interviews.

Patients will complete baseline geriatric assessments and a 30-45-minute cognitive test, and both will be reassessed in 3 months intervals. The geriatric assessment is primarily patient-reported surveys and involves a multi-domain evaluation of a patient's functional status (i.e., their ability to live independently at home and in the community), co-morbid medical conditions, cognition, psychological status, social functioning and support, medications, and nutritional status. Care Partners will be asked to complete baseline surveys that will also assess their well-being and ability to function at home.

To provide a more comprehensive understanding of the myeloma-related experiences a subset of patients and their care partners will be asked to participate in a baseline interview repeated over time to understand how the disease and its treatments shape the experiences.

Duration of Subject Participation: 6 months

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following inclusion criteria to participate in this study:

1. Aged ≥55
2. New myeloma diagnosis as defined by the International Myeloma Working Group, does not have another non-myeloma plasma cell disorder such as POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal plasma cell disorder, skin changes) or amyloidosis.
3. Starting systemic treatment.
4. Able to understand and speak in English.
5. Able to provide informed consent to participate.

Care Partners must meet the following inclusion criteria to participate in this study

1. Aged ≥18.
2. Able to understand and speak in English.
3. Able to provide informed consent to participate.
4. Be a care partner for a patient with multiple myeloma and is also enrolled in the assessment portion of this study.
5. Willing and able to participate in semi-structured interviews.

Exclusion Criteria:

1. All participants meeting any of the following exclusion criteria at enrollment will be excluded from the study: Inability to read and speak English.
2. Dementia altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study has two different population groups: A. Forty subjects with newly diagnosed multiple myeloma did not receive treatment yet., B. Thirty care partners of the subjects with newly diagnosed multiple myeloma did not receive treatment yet.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Trajectories of cognitive functions NIHTB-CB | Up to 6 months
  Standardized National Institutes of Health Toolbox Cognition Battery (objective) (NIHTB-CB) will be used for the measure of cognitive function. The NIHTB-CB contains 7 computer-based instruments assessing 5 cognitive sub-domains: Language, Executive Function, Episodic Memory, Processing Speed, and Working Memory. The Composite Score is calculated using all subsets. Higher score =better level of cognitive functions.
Trajectories of cognitive functions PROMIS | Up to 6 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v2.0 - Cognitive function 8a (subjective) scores will be combined for an overall measure of cognitive function. PROMIS Short Form v2.0- Cognitive function 8a is a participant reported measure of cognitive function. There are 8 questions, with a possible raw score of 8 to 40, then converted into a T-score for each participant. T-scores lower below 50 indicate a lower than average cognitive performance.
Trajectories of HRQoL cognitive functions | Up to 6 months
  The European Organization for Research and Treatment of Cancer Quality-of-Life questionnaire (EORTC QLQ-C30) will be used to measure the changes in quality of life. EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. EORTC QLQ-C30 includes functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting), and other (dyspnea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties). Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score=better level of physical functioning.
Trajectories of physical function measured by ADLs | Up to 6 months
  The physical function will be measured using participant-reported activities of daily living (ADLs) as bath, dress, toilet, transfer bed to chair, maintain continence and feed. The score ranges from 0-6 with an increasing score indicating loss of independence/function.
Trajectories of physical function measured by IADLS | Up to 6 months
  The physical function will be measured using Older Americans Resources and Services (OARS) instrumental activities of daily living (IADLS). Participants are asked to self-report their ability to engage in the following activities of daily living: bathe, dress, feed, toilet, maintain continence, transfer from bed to chair, use the telephone, shop, prepare food, housekeeping, laundry, take medications, manage finances, use transportation. The score ranges from 0-8 with an increasing score indicating loss of independence/function.
Trajectories of physical function measured by Gait speed | Up to 6 months
  The physical function will be measured using gait speed. Gait speed is measured by having participants walk at their normal pace at a distance of 4 meters. The slower the gait speed the more likely an individual is likely to be impaired functionally.

SECONDARY OUTCOMES:
Predictors of changes in cognitive function | Up to 6 months
  Multivariable regression modelling will be used to examine whether or not the following participant-reported socio-demographics factors (age, race, sex, education, income, community social vulnerability) and geriatric conditions (medical comorbidities, depression, anxiety, lack of social support) can predict those most likely to experience changes in cognitive function over a 6- month period.
Predictors of changes in physical function | Up to 6 months
  Multivariable regression modelling will be used to examine whether or not the following participant-reported socio-demographics factors (age, race, sex, education, income, community social vulnerability) and geriatric conditions (medical comorbidities, depression, anxiety, lack of social support) can predict those most likely to experience changes in physical function (ADLS, IADLS, gait speed) over a 6-month period.
Predictors of changes in quality of life | Up to 6 months
  Multivariable regression modeling will be used to examine whether or not the following participant-reported socio-demographics factors (age, race, sex, education, income, community social vulnerability) and geriatric conditions (medical comorbidities, depression, anxiety, lack of social support) can predict those most likely to experience changes in quality of life level based on the European Organization for Research and Treatment of Cancer Quality-of-Life questionnaire (EORTC QLQ-C30) scores, over 6- month period. Higher score=better level of physical functioning.
Gain a complete understanding of the challenges patients and care partners living with multiple myeloma face | Up to 6 months
  Multiple myeloma and its associated treatments shape functional capacity, quality of life, and the overall illness experience in adults with multiple myeloma and their care partners will be evaluated using semi-structured interviews. Furthermore, changes between baseline, and at 3 months after treatment starts will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Shakira Grant, MBBS, Principal Investigator — Lineberger CCC, Center for Aging and Health, The University of North Carolina Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — https://unclineberger.org/patientcare/clinical-trials/